CLINICAL TRIAL: NCT03278847
Title: Optimising Newborn Nutrition During Therapeutic Hypothermia: an Observational Study Using Routinely Collected Data
Brief Title: Optimising Newborn Nutrition During Therapeutic Hypothermia.
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: University of Nottingham (Other); Bliss Charity (Other)
Responsible Party: Sponsor
Other Study IDs: 17IC4064; 16/79/03 (Other Grant/Funding Number: National Institute for Health Research (NIHR) HTA); 17/EM/0307 (Other: United Kingdom Health Research Authority)
Record Dates: First submitted 2017-08-23; First posted 2017-09-12 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2022-11

CONDITIONS: Infant, Newborn; Asphyxia Neonatorum; Hypothermia, Induced; Parenteral Nutrition; Infant Nutrition; Necrotizing Enterocolitis; Neonatal Sepsis
Keywords: NNRD; matching; propensity score
MeSH Terms: conditions — Asphyxia Neonatorum; Hypothermia; Hyperphagia; Enterocolitis, Necrotizing; Neonatal Sepsis | interventions — Milk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Enteral nutrition comparison: This comparison refers to differences in enteral nutrition during therapeutic hypothermia
  Interventions: Dietary Supplement: Received enteral (milk) feeds during therapeutic hypothermia; Dietary Supplement: Enteral (milk) feeds withheld during therapeutic hypothermia
- Parenteral nutrition comparison: This comparison refers to differences in parenteral nutrition during therapeutic hypothermia
  Interventions: Dietary Supplement: Received parenteral nutrition during therapeutic hypothermia; Dietary Supplement: Did not receive parenteral nutrition during therapeutic hypothermia

INTERVENTIONS:
Dietary Supplement: Received enteral (milk) feeds during therapeutic hypothermia — In the enteral component of nutrition, the health technology to be assessed is the gradual introduction of enteral (milk) feeds during therapeutic hypothermia:
  * Included in this is any type of milk (e.g. expressed maternal breast milk, expressed donor breast milk and artificial formula)
  * This health technology includes different routes of administering enteral feeds such as nasogastric tube (gavage feeding) and bottle
  * This health technology also includes different rates of increasing enteral feeds (for example by 15ml/kg/day, by 30ml/kg/day or faster)
  Groups: Enteral nutrition comparison
Dietary Supplement: Enteral (milk) feeds withheld during therapeutic hypothermia — Withholding enteral feeds (keeping a baby nil per os) for the duration of hypothermia.
  Groups: Enteral nutrition comparison
Dietary Supplement: Received parenteral nutrition during therapeutic hypothermia — In the parenteral component, the health technology being assessed is administration of parenteral nutrition during therapeutic hypothermia:
  * Included in this are different compositions of parenteral nutrition (for example standard, pre-prepared bags of nutrition and individually tailored parenteral nutrition)
  * This health technology includes different routes of administration of parenteral nutrition such as via a peripheral intravenous cannula, percutaneous central venous catheter ('long line') or umbilical venous catheter.
  * This health technology also includes different volumes of parenteral nutrition (e.g. 40ml/kg/day, 60ml/kg/day or greater).
  Groups: Parenteral nutrition comparison
Dietary Supplement: Did not receive parenteral nutrition during therapeutic hypothermia — Received standard intravenous fluids (10% dextrose with additional electrolytes added where required) for the duration of hypothermia.
  Groups: Parenteral nutrition comparison

SUMMARY:
The overarching aim of this project is to determine the optimum enteral and parenteral nutrition strategy for newborns with Hypoxic Ischaemic Encephalopathy (HIE) during and after therapeutic hypothermia. To do this the investigators will perform two primary comparisons:

1. ENTERAL: to determine whether any enteral (milk) feeding, when compared to withholding enteral feeding (no milk), during therapeutic hypothermia, is associated with a difference in the incidence of necrotising enterocolitis.
2. PARENTERAL: to determine whether provision of intravenous dextrose, when compared to provision of parenteral nutrition, during therapeutic hypothermia, is associated with a difference in the incidence of blood stream infection.

The investigators will use de-identified data held in an established research database called the National Neonatal Research Database (NNRD) and we will use the potential outcomes framework with application of propensity scoring to define matched subgroups for comparison.

DETAILED DESCRIPTION:
Every year about 1200 babies in England, Wales and Scotland suffer from a lack of oxygen around birth which can lead to long-term brain injury or death. This is called Hypoxic Ischaemic Encephalopathy (HIE). Research has shown that cooling babies with HIE by a few degrees for the first 3 days protects the brain; all babies with moderate or severe HIE in the UK are treated with therapeutic hypothermia (cooling).

Doctors do not know how best to care for babies while they are cooled. A key question is "how to provide nutrition to babies during cooling". There are two main parts to this question, milk feeds ("enteral" nutrition) and intravenous nutrition ("parenteral" nutrition). Doctors don't know how best to provide either milk or intravenous nutrition to cooled babies.

* MILK FEEDS: Some neonatal units in the UK carefully feed babies (usually with maternal breast milk) while they are cooled. This avoids intravenous lines and is believed to help them feed and go home earlier. Other neonatal units do not feed cooled babies because they worry about a condition called necrotising enterocolitis (a devastating and often fatal disease) which might be more common with feeding.
* INTRAVENOUS NUTRITION: All cooled babies need intravenous fluid (even when milk feeds are given it takes several days before enough fluid can be given this way). Some neonatal units give babies intravenous nutrition (which contains fat, protein, carbohydrate, vitamins and minerals) as this may improve growth and recovery. Other neonatal units only give intravenous dextrose with simple salts because of concerns that intravenous nutrition leads to more infections. This study will compare these different ways of providing nutrition. It will use a research database called the National Neonatal Research Database (NNRD). In England, Scotland and Wales doctors and nurses looking after babies in neonatal care (including all cooled babies) use an Electronic Health Record system. Data from this system are anonymised (no baby can be identified) and form the NNRD, so the NNRD holds data from all babies who have been looked after on NHS neonatal units.

The investigators have worked closely with parents and charities in developing the NNRD. The investigators will use the NNRD to study all term babies who received cooling in England, Scotland and Wales since 2008. The investigators will compare the milk feeding and intravenous nutrition they receive.

* MILK FEEDING: The investigators will compare babies who are fed milk while cooled with those that are not fed any milk. The investigator's main goal is to establish whether there is any difference in rates of necrotising enterocolitis.
* INTRAVENOUS NUTRITION: The investigators will compare babies who get intravenous nutrition with those that only get intravenous dextrose. The main difference we are looking for is in the rate of infection. The investigators will also study how many babies die, how long they stay in neonatal care, how soon breastfeeding starts and many are breastfed when they go home.

The investigators will apply a statistical approach called "potential outcomes framework" in which babies are matched in each group (e.g. babies who are fed and those who are not fed) as closely as possible. This will ensure that any difference in outcomes is due to the different nutritional treatments and not due to background differences or other confounders (like how sick a baby is).

The results from this study will help to ensure that babies who need to be cooled for HIE receive the best and safest nutrition in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Received neonatal care at a unit that is part of the UK Neonatal Collaborative; this includes all NHS neonatal units in England, Scotland and Wales
2. Recorded gestational age at birth ≥36 weeks
3. Recorded as receiving therapeutic hypothermia for 72 hours or died during therapeutic hypothermia

Exclusion Criteria:

1. Infants with missing data for principal background and outcome variables.

Max Age: 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants born at 36 gestational weeks or later who received therapeutic hypothermia for Hypoxic Ischaemic Encephalopathy (HIE) for least 72 hours, or who died during therapeutic hypothermia.
Sampling Method: Non-Probability Sample
Enrollment: 6030 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Gale, MBBS, PhD, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Chelsea and Westminster Hospital and NHS Foundation Trust, London
  - Imperial College London, Chelsea and Westminster Hospital campus, London

IPD SHARING:
Plan to Share IPD: Yes
All study data will be extracted from the National Neonatal Research Database (NNRD). The NNRD has been created through the collaborative efforts of neonatal services across the country to be a national resource. The NNRD is maintained and managed at the Neonatal Data Analysis Unit (NDAU) at Imperial College London and Chelsea and Westminster NHS Foundation Trust.
  Researchers, clinicians, managers, commissioners, and others are welcome and encouraged to utilise the NNRD.
Supporting Information: Study Protocol, CSR
Time Frame: The NNRD holds data from 2007 to present.
Access Criteria: Access criteria and guidance is found at the URL below
URL: https://www.imperial.ac.uk/neonatal-data-analysis-unit/neonatal-data-analysis-unit/utilising-the-national-neonatal-research-database/

REFERENCES:
- [Background] Battersby C, Longford N, Patel M, Selby E, Ojha S, Dorling J, Gale C. Study protocol: optimising newborn nutrition during and after neonatal therapeutic hypothermia in the United Kingdom: observational study of routinely collected data using propensity matching. BMJ Open. 2018 Oct 23;8(10):e026739. doi: 10.1136/bmjopen-2018-026739. PMID 30355795
- [Background] Gale C, Jeyakumaran D, Longford N, Battersby C, Ojha S, Oughham K, Dorling J. Administration of parenteral nutrition during therapeutic hypothermia: a population level observational study using routinely collected data held in the National Neonatal Research Database. Arch Dis Child Fetal Neonatal Ed. 2021 Nov;106(6):608-613. doi: 10.1136/archdischild-2020-321299. Epub 2021 May 5. PMID 33952628
- [Result] Gale C, Longford NT, Jeyakumaran D, Ougham K, Battersby C, Ojha S, Dorling J. Feeding during neonatal therapeutic hypothermia, assessed using routinely collected National Neonatal Research Database data: a retrospective, UK population-based cohort study. Lancet Child Adolesc Health. 2021 Jun;5(6):408-416. doi: 10.1016/S2352-4642(21)00026-2. Epub 2021 Apr 21. PMID 33891879
- [Result] Gale C, Jeyakumaran D, Battersby C, Ougham K, Ojha S, Culshaw L, Selby E, Dorling J, Longford N. Nutritional management in newborn babies receiving therapeutic hypothermia: two retrospective observational studies using propensity score matching. Health Technol Assess. 2021 Jun;25(36):1-106. doi: 10.3310/hta25360. PMID 34096500

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an observational study. 6030 babies were included in the overall study cohort and from this two pairs of matched groups were formed to examine the impact of enteral feeding during therapeutic hypothermia (two matched groups of 1618) and of parenteral nutrition during therapeutic hypothermia (two matched groups of 1240).
Groups:
- Received Enteral (Milk) Feeds During Therapeutic Hypothermia: The gradual introduction of enteral (milk) feeds during therapeutic hypothermia:
  * Included in this is any type of milk (e.g. expressed maternal breast milk, expressed donor breast milk and artificial formula)
  * This health technology includes different routes of administering enteral feeds such as nasogastric tube (gavage feeding) and bottle
  * This health technology also includes different rates of increasing enteral feeds (for example by 15ml/kg/day, by 30ml/kg/day or faster)
- Received Parenteral Nutrition During Therapeutic Hypothermia:: Administration of parenteral nutrition during therapeutic hypothermia:
  * Included in this are different compositions of parenteral nutrition (for example standard, pre-prepared bags of nutrition and individually tailored parenteral nutrition)
  * This health technology includes different routes of administration of parenteral nutrition such as via a peripheral intravenous cannula, percutaneous central venous catheter ('long line') or umbilical venous catheter.
  * This health technology also includes different volumes of parenteral nutrition (e.g. 40ml/kg/day, 60ml/kg/day or greater).
Period: Overall Study
Arm/Group | Received Enteral (Milk) Feeds During Therapeutic Hypothermia | Enteral (Milk) Feeds Withheld During Therapeutic Hypothermia | Received Parenteral Nutrition During Therapeutic Hypothermia: | Did Not Receive Parenteral Nutrition During Therapeutic Hypothermia
Started | 1618 | 1618 | 1240 | 1240
Completed | 1618 | 1618 | 1240 | 1240
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Received Enteral (Milk) Feeds During Therapeutic Hypothermia | Enteral (Milk) Feeds Withheld During Therapeutic Hypothermia | Received Parenteral Nutrition During Therapeutic Hypothermia: | Did Not Receive Parenteral Nutrition During Therapeutic Hypothermia | Total
Number analyzed (Participants) | 1618 | 1618 | 1240 | 1240 | 5716
Age, Customized [Mean (Standard Deviation); unit: Weeks] — Gestation at birth in weeks Population: This is a factorial study where the same group of babies were included in enteral and parenteral nutrition analyses
  Weeks
    Enteral feeding: number analyzed (Participants) | 1618 | 1618 | 0 | 0 | 3236
    Enteral feeding | 39.5 (1.5) | 39.5 (1.5) |  |  | 39.5 (1.5)
    Parenteral feeding: number analyzed (Participants) | 0 | 0 | 1240 | 1240 | 2480
    Parenteral feeding |  |  | 39.4 (1.6) | 39.4 (1.6) | 39.4 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This is a factorial study where the same group of babies were included in enteral and parenteral nutrition analyses
  Participants
    Enteral feeding: number analyzed (Participants) | 1618 | 1618 | 0 | 0 | 3236
    Enteral feeding: Female | 715 | 715 | 0 | 0 | 1430
    Enteral feeding: Male | 903 | 903 | 0 | 0 | 1806
    Parenteral nutrition: number analyzed (Participants) | 0 | 0 | 1240 | 1240 | 2480
    Parenteral nutrition: Female | 0 | 0 | 576 | 588 | 1164
    Parenteral nutrition: Male | 0 | 0 | 664 | 652 | 1316
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: This is a factorial study where the same group of babies were included in enteral and parenteral nutrition analyses
  Participants
    Enteral feeding - White: number analyzed (Participants) | 1618 | 1618 | 0 | 0 | 3236
    Enteral feeding - White | 1040 | 1041 |  |  | 2081
    Enteral feeding - Asian or mixed Asian: number analyzed (Participants) | 1618 | 1618 | 0 | 0 | 3236
    Enteral feeding - Asian or mixed Asian | 169 | 174 |  |  | 343
    Enteral feeding - Black or mixed black African: number analyzed (Participants) | 1618 | 1618 | 0 | 0 | 3236
    Enteral feeding - Black or mixed black African | 103 | 99 |  |  | 202
    Enteral feeding - Other and missing: number analyzed (Participants) | 1618 | 1618 | 0 | 0 | 3236
    Enteral feeding - Other and missing | 306 | 304 |  |  | 610
    Parenteral nutrition - White: number analyzed (Participants) | 0 | 0 | 1240 | 1240 | 2480
    Parenteral nutrition - White |  |  | 991 | 1002 | 1993
    Parenteral nutrition - Asian or Mixed Asian: number analyzed (Participants) | 0 | 0 | 1240 | 1240 | 2480
    Parenteral nutrition - Asian or Mixed Asian |  |  | 93 | 98 | 191
    Parenteral nutrition - Black or mixed black African: number analyzed (Participants) | 0 | 0 | 1240 | 1240 | 2480
    Parenteral nutrition - Black or mixed black African |  |  | 62 | 53 | 115
    Parenteral nutrition - Other and missing: number analyzed (Participants) | 0 | 0 | 1240 | 1240 | 2480
    Parenteral nutrition - Other and missing |  |  | 94 | 86 | 180
Region of Enrollment [Number; unit: participants] — Population: This is a factorial study where the same group of babies were included in enteral and parenteral nutrition analyses
  participants
    United Kingdom: number analyzed (Participants) | 1618 | 1618 | 0 | 0 | 3236
    United Kingdom | 1618 | 1618 |  |  | 3236
Region of Enrollment [Number; unit: participants]
  United Kingdom | 0 | 0 | 1240 | 1240 | 2480
Cord pH <6.9 [Count of Participants; unit: Participants] — Population: This is a factorial study where the same babies are included in both enteral and parenteral analyses
  Participants
    Enteral feeding: number analyzed (Participants) | 1618 | 1618 | 0 | 0 | 3236
    Enteral feeding | 368 | 368 |  |  | 736
    Parenteral nutrition: number analyzed (Participants) | 0 | 0 | 1240 | 1240 | 2480
    Parenteral nutrition |  |  | 280 | 280 | 560
Apgar score 0 or 1 at 5 minutes [Count of Participants; unit: Participants] — Population: This is a factorial study where the same babies are included in both enteral and parenteral analyses
  Participants
    Enteral feeding: number analyzed (Participants) | 1618 | 1618 | 0 | 0 | 3236
    Enteral feeding | 678 | 720 |  |  | 1398
    Parenteral nutrition: number analyzed (Participants) | 0 | 0 | 1240 | 1240 | 2480
    Parenteral nutrition |  |  | 562 | 553 | 1115
Treatment with inotropes on day of admission [Count of Participants; unit: Participants] — Population: This is a factorial study and the same babies are included in both enteral and parenteral analyses
  Participants
    Enteral feeding: number analyzed (Participants) | 1618 | 1618 | 0 | 0 | 3236
    Enteral feeding | 288 | 295 |  |  | 583
    Parenteral nutrition: number analyzed (Participants) | 0 | 0 | 1240 | 1240 | 2480
    Parenteral nutrition |  |  | 287 | 295 | 582

OUTCOME MEASURES:

1. Primary Outcome: Necrotising Enterocolitis - for the Enteral Nutrition Comparison
Description: Defined according to the case definition of Battersby et al., 2017, JAMA Pediatrics
Time Frame: From date of birth until date of final neonatal unit discharge, assessed up to 1 year
Population: NA indicates <5 where the cell value is withheld to avoid identifying participants
Measure: Count of Participants; unit: Participants
Arm/Group | Received Enteral (Milk) Feeds During Therapeutic Hypothermia | Enteral (Milk) Feeds Withheld During Therapeutic Hypothermia | Received Parenteral Nutrition During Therapeutic Hypothermia: | Did Not Receive Parenteral Nutrition During Therapeutic Hypothermia
Number analyzed (Participants) | 1618 | 1618 | 1240 | 1240
Participants | NA — NA indicates <5 where the cell value is withheld to avoid identifying participants | NA — NA indicates <5 where the cell value is withheld to avoid identifying participants | NA — NA indicates <5 where the cell value is withheld to avoid identifying participants | 7

2. Primary Outcome: Blood Stream Infection - for the Parenteral Nutrition Comparison
Description: defined according to the Healthcare Quality Improvement Partnership (HQIP) National Neonatal Audit Programme (NNAP) case definition: pure growth of a recognised pathogen from a normally sterile site
Time Frame: From date of birth until date of final neonatal unit discharge, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Received Enteral (Milk) Feeds During Therapeutic Hypothermia | Enteral (Milk) Feeds Withheld During Therapeutic Hypothermia | Received Parenteral Nutrition During Therapeutic Hypothermia: | Did Not Receive Parenteral Nutrition During Therapeutic Hypothermia
Number analyzed (Participants) | 1618 | 1618 | 1240 | 1240
Participants | NA — NA indicates <5 where the cell value is withheld to avoid identifying participants | 8 | 11 | NA — NA indicates <5 where the cell value is withheld to avoid identifying participants

3. Secondary Outcome: Survival
Description: Survival at neonatal unit discharge
Time Frame: From date of birth until date of final neonatal unit discharge, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Received Enteral (Milk) Feeds During Therapeutic Hypothermia | Enteral (Milk) Feeds Withheld During Therapeutic Hypothermia | Received Parenteral Nutrition During Therapeutic Hypothermia: | Did Not Receive Parenteral Nutrition During Therapeutic Hypothermia
Number analyzed (Participants) | 1618 | 1618 | 1240 | 1240
Participants | 1552 | 1465 | 1154 | 1116

4. Secondary Outcome: Length of Stay
Description: Number of days between first neonatal unit admission and final neonatal unit discharge for surviving infants
Time Frame: From date of birth until date of final neonatal unit discharge, assessed up to 1 year
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Received Enteral (Milk) Feeds During Therapeutic Hypothermia | Enteral (Milk) Feeds Withheld During Therapeutic Hypothermia | Received Parenteral Nutrition During Therapeutic Hypothermia: | Did Not Receive Parenteral Nutrition During Therapeutic Hypothermia
Number analyzed (Participants) | 1618 | 1618 | 1240 | 1240
Days | 12.7 [12.0 to 13.3] | 14.8 [14.2 to 15.5] | 15.0 [14.1 to 15.8] | 14.1 [13.6 to 14.7]

5. Secondary Outcome: Breastfeeding
Description: Any breastfeeding (suckling at the breast) at discharge
Time Frame: At the point of final discharge from neonatal care, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Received Enteral (Milk) Feeds During Therapeutic Hypothermia | Enteral (Milk) Feeds Withheld During Therapeutic Hypothermia | Received Parenteral Nutrition During Therapeutic Hypothermia: | Did Not Receive Parenteral Nutrition During Therapeutic Hypothermia
Number analyzed (Participants) | 1618 | 1618 | 1240 | 1240
Participants | 883 | 752 | 575 | 582

6. Secondary Outcome: Hypoglycaemia
Description: Any diagnosis of hypoglycaemia recorded after therapeutic hypothermia is commenced and before the final neonatal unit discharge
Time Frame: From date of birth until date of final neonatal unit discharge, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Received Enteral (Milk) Feeds During Therapeutic Hypothermia | Enteral (Milk) Feeds Withheld During Therapeutic Hypothermia | Received Parenteral Nutrition During Therapeutic Hypothermia: | Did Not Receive Parenteral Nutrition During Therapeutic Hypothermia
Number analyzed (Participants) | 1618 | 1618 | 1240 | 1240
Participants | 293 | 269 | 212 | 235

7. Secondary Outcome: Duration of Central Venous Line
Description: The number of days until an infant is recorded as not having a central venous line
Time Frame: From date of birth until date of final neonatal unit discharge, assessed up to 1 year
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Received Enteral (Milk) Feeds During Therapeutic Hypothermia | Enteral (Milk) Feeds Withheld During Therapeutic Hypothermia | Received Parenteral Nutrition During Therapeutic Hypothermia: | Did Not Receive Parenteral Nutrition During Therapeutic Hypothermia
Number analyzed (Participants) | 1618 | 1618 | 1240 | 1240
Days | 4.3 [4.1 to 4.5] | 5.5 [5.3 to 5.7] | 6 [5.7 to 6.3] | 5.1 [5 to 5.3]

8. Secondary Outcome: Growth
Description: Weight for post-menstrual age standard deviation score at final neonatal unit discharge.
  Standard deviation score, higher score means higher growth (higher weight for gestational age)
Time Frame: From date of birth until date of final neonatal unit discharge, assessed up to 1 year
Measure: Mean (95% Confidence Interval); unit: Standard deviation score
Arm/Group | Received Enteral (Milk) Feeds During Therapeutic Hypothermia | Enteral (Milk) Feeds Withheld During Therapeutic Hypothermia | Received Parenteral Nutrition During Therapeutic Hypothermia: | Did Not Receive Parenteral Nutrition During Therapeutic Hypothermia
Number analyzed (Participants) | 1618 | 1618 | 1240 | 1240
Standard deviation score | -0.54 [-0.59 to -0.48] | -0.6 [-0.65 to -0.55] | -0.65 [-0.71 to -0.58] | -0.66 [-0.71 to -0.61]

ADVERSE EVENTS:
Time Frame: Until end of neonatal unit stay
Arm/Group | Received Enteral (Milk) Feeds During Therapeutic Hypothermia | Enteral (Milk) Feeds Withheld During Therapeutic Hypothermia | Received Parenteral Nutrition During Therapeutic Hypothermia: | Did Not Receive Parenteral Nutrition During Therapeutic Hypothermia
All-Cause Mortality (participants affected / at risk) | 66/1618 | 153/1618 | 86/1240 | 124/1240
Serious Adverse Events (participants affected / at risk) | 0/1618 | 0/1618 | 0/1240 | 0/1240
Other Adverse Events (participants affected / at risk) | 0/1618 | 0/1618 | 0/1240 | 0/1240

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT03278847/Prot_SAP_000.pdf